CLINICAL TRIAL: NCT06305741
Title: Managing Anxiety From Cancer (MAC): Evaluation of a Tailored Anxiety Intervention for Latino Older Adults With Cancer and Their Caregivers
Brief Title: A Study of an Anxiety Intervention for Latino/Latina/Hispanic Older Adults With Cancer and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-060
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Cancer Patients; Care Givers
Keywords: Anxiety Intervention; Latino caregivers; 24-060

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Latino caregivers and the Latino older adults with cancer (OACs) (Experimental): The intervention, MAC, is a seven-session (45- 60 minutes per session) psychotherapy intervention delivered via videoconference and/or telephone by licensed social workers. All sessions will be audio-recorded. MAC content, structure, and length are consistent with core components of cognitive behavioral therapy (CBT) (Freeman, 2004).
  Interventions: Other: Managing Anxiety from Cancer (MAC)

INTERVENTIONS:
Other: Managing Anxiety from Cancer (MAC) — The intervention, MAC, is a seven-session (45-60 minutes per session) psychotherapy intervention delivered via videoconference.
  and/or telephone by licensed social workers

SUMMARY:
The purpose of this study is to find out if an anxiety treatment program is practical and effective for Latino older adults with cancer (OACs) and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

Older Adults with Cancer (OAC)

* As per medical record or self-report, is currently age 65 years or older
* As per medical record or self-report, currently receiving active cancer treatment OR is within eighteen months of completing active treatment which includes surgery, chemotherapy, radiation, and immunotherapy.
* As per self-report, identifies as Latino and/or Hispanic Ethnicity
* Per self-report, has a primary informal caregiver (as defined by an unpaid individual who provides the patient with emotional, physical, and/or practical support) age 40 or older who is willing and able to participate in the study ; if a patient does not have a primary informal caregiver or if the caregiver does not or cannot participate, but meets all other inclusion criteria they will be allowed to enroll in the study
* Scores ≥6 on the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS)
* Per self-report, fluent in English and/or Spanish** ** Language verification: Prior to enrollment, patients will be asked the following two questions by a Clinical Research Coordinator (CRC) to verify language fluency necessary for participation in the study:

  1. How well do you speak English and/or Spanish? (must respond "very well" or "well" when given the choices of Very well, Well, Not well, Not at all, Don't know, or Refused)
  2. What is your preferred language for healthcare? (must respond English and/or Spanish)

Caregiver

* Per OAC report, is primary informal caregiver (as defined by an unpaid individual who provides the patient with emotional, physical, and/or practical support) for the eligible OAC patient
* As per self-report, is age 40 years or older
* Per self-report, fluent in English and/or Spanish** ** Language verification: Prior to enrollment, patients will be asked the following two questions by a Clinical Research Coordinator (CRC) to verify language fluency necessary for participation in the study:

  1. How well do you speak English and/or Spanish? (must respond "very well" or "well" when given the choices of Very well, Well, Not well, Not at all, Don't know, or Refused)
  2. What is your preferred language for healthcare? (must respond English and/or Spanish)

Exclusion Criteria:

OAC

* As per medical record or self-report, currently receiving psychotherapy
* As per medical record or self-report, taking psychotropic medications for < 8 weeks prior to MAC Session 1 and/or anticipates changing their medication during the study
* As per medical record or self-report, currently being treated for schizophrenia, substance use or dependence, and/or bi-polar disorder
* Severely cognitively impaired as demonstrated by Blessed Orientation Memory Concentration score ≥ 9
* Per research staff judgment and/or self-report, too ill or weak to complete study procedures
* Per medical record or self-report, receiving hospice care at the time of enrollment

Caregiver

* As per self-report, currently receiving psychotherapy
* As per self-report, taking psychotropic medications for < 8 weeks prior to MAC Session 1 and/or anticipates changing their medication during the study
* As per self-report, currently being treated for schizophrenia, substance use or dependence, and/or bi-polar disorder
* Severely cognitively impaired as demonstrated by Blessed Orientation Memory Concentration score ≥ 11
* Per research staff judgment and/or self-report, too ill or weak to complete study procedures

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
percentage of participants to complete all study procedures | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kelly McConnell, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm